CLINICAL TRIAL: NCT03581149
Title: Tolerability and Efficacy of Low-Volume Sodium Picosulfate/Magnesium Citrate Versus 2L Polyethylene Glycol/Ascorbic Acid in Patients With Ulcerative Colitis Undergoing Colonoscopy: A Randomized Controlled Trial
Brief Title: Tolerability and Efficacy of Sodium Picosulfate/Magnesium Citrate Versus PEG/Ascorbic Acid in Ulcerative Colitis Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Ala'a Sharara, MD, Professor, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: BIO-2017-0434
Record Dates: First submitted 2018-03-27; First posted 2018-07-10 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — picosulfate sodium; Polyethylene Glycols; Ascorbic Acid; MoviPrep

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Citrafleet® (Active Comparator): Patients will receive sodium picosulfate/magnesium citrate (Citrafleet®) solution with an instruction leaflet.
  Interventions: Drug: Sodium Picosulfate/Magnesium Citrate Laxative
- MoviPrep® (Active Comparator): Patients will receive 2L polyethylene glycol + ascorbic acid (MoviPrep®) solution with an instruction leaflet.
  Interventions: Drug: 2L polyethylene glycol/ascorbic acid

INTERVENTIONS:
Drug: Sodium Picosulfate/Magnesium Citrate Laxative — ● First arm: Patients will receive sodium picosulfate/magnesium citrate (Citrafleet®) solution with an instruction leaflet.
  Other Names: (Citrafleet®)
  Arms: Citrafleet®
Drug: 2L polyethylene glycol/ascorbic acid — * First arm: Patients will receive sodium picosulfate/magnesium citrate (Citrafleet®) solution with an instruction leaflet.
  * Second arm: Patients will receive 2L polyethylene glycol + ascorbic acid (MoviPrep®) solution with an instruction leaflet.
  Other Names: (MoviPrep®)
  Arms: MoviPrep®

SUMMARY:
Ulcerative colitis is a chronic condition that results in the inflammation of the colon and rectum. Patients suspected to have ulcerative colitis are diagnosed via colonoscopy. Moreover, colonoscopy is considered to be the preferred procedure for assessing the activity and extent of the disease, as well as monitoring treatment response and development of lesions. Therefore, optimal performance and visualization of mucosal lesions via adequate bowel preparation is essential in such patients. In addition, the nature of the disease and the need for multiple colonoscopies throughout a patient's lifetime makes compliance to repeated procedures difficult.

It is well known that colonoscopy preparations are generally poorly tolerated, disliked and, consequently serve as an additional burden on patients.Polyethylene glycol (PEG), despite being the golden standard, is not very well tolerated. Inadequate bowel preparations are associated with cancelled procedures, prolonged procedure time, incomplete examination, increased cost and possibly complications, physician frustration and patient anxiety, but most importantly, with missed pathology. A good bowel preparation would need a solution with reasonable volume, acceptable taste, minimal diet restrictions, and easy-to-follow instructions. The strict need for adherence to drinking a relatively large volume of solution preparation may result in poor compliance.

Despite the emergence of several types of low volume preparations, the evidence on the use of such solutions remains sparse. This is especially true in terms of patients' tolerability to the solution, and its relation with adequate bowel preparation during colonoscopy.

The investigator's aim is to assess how small volume preparations such as sodium picosulfate/magnesium citrate (Citrafleet®) enhance participants tolerability to the solution, compliance, and adequacy of bowel preparations when compared to 2L polyethylene glycol + ascorbic acid (MoviPrep®) in patients with Ulcerative Colitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Ulcerative Colitis
* Patients undergoing elective outpatient colonoscopy
* Patients consenting to the study

Exclusion Criteria:

* Age less than 18 years
* Pregnant or lactating women
* Significant gastroparesis
* Gastric outlet obstruction
* Ileus
* Known or suspected bowel obstruction or perforation
* Phenylketonuria
* Toxic colitis or megacolon
* Having a stoma
* Compromised swallowing reflex or mental status
* Psychiatric disease or known or suspected poor compliance
* Severe chronic renal failure (creatinine clearance <30 mL/minute)
* Severe congestive heart failure (New York Heart Association [NYHA] class III or IV)
* Dehydration
* Laxative use or dependency
* Chronic constipation (<3 spontaneous bm/week)
* Uncontrolled hypertension (systolic blood pressure ≥170 mm Hg, diastolic blood pressure ≥100 mm Hg)
* Prior colon resection
* Age above 65 years
* Profusely bleeding patients with severe UC

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2018-03-26 (Actual); Primary Completion 2020-07-26 (Estimated); Study Completion 2020-07-26 (Estimated)

PRIMARY OUTCOMES:
Tolerability of the preparation as assessed by a Likert-type scale | 1 year
  Patients will answer a data collection sheet with questions regarding their ability to tolerate the preparation without difficulty. We are using a Likert-type scale from 1 to 5, 1 being completely intolerable and 5 being very easily tolerated.

SECONDARY OUTCOMES:
Quality of the preparation as assessed by the Modified Aronchick scale. | 1 year
  A data collection sheet will be handed to the blinded endoscopist to answer questions related to the quality of the preparation. A description ranging from Poor to Excellent is assigned to the quality of the prepped colon.
  Poor - Re-preparation required; large amount of fecal residue precludes a complete examination
  Inadequate - Inadequate but examination completed; enough feces or turbid fluid to prevent a reliable examination; less than 90%mucosa seen
  Fair - Moderate amount of stool that can be cleared with suctioning permitting adequate evaluation of entire colonic mucosa; more than 90% mucosa seen
  Good - Small amount of turbid fluid without feces not interfering with examination; more than 90% mucosa seen
  Excellent - Small amount of clear liquid with clear mucosa seen; more than 95% mucosa seen
Quality of the preparation as assessed by the Boston Bowel Preparation Scale. | 1 year
  A data collection sheet will be handed to the blinded endoscopist to answer questions related to the quality of the preparation. A score ranging from 0 to 3 is assigned to each of the three segments of the colon: Right colon, Mid colon and Left colon. The scores are calculated as follows:
  0 = Unprepared colon segment with mucosa not seen due to solid stool that cannot be cleared.
  1. = Portion of mucosa of the colon segment seen, but other areas of the colon segment not well seen due to staining, residual stool and/or opaque liquid.
  2. = Minor amount of residual staining, small fragments of stool and/or opaque liquid, but mucosa of colon segment seen well.
  3. = Entire mucosa of colon segment seen well with no residual staining, small fragments of stool or opaque liquid.
Assessment of adherence to protocol | 1 year
  Patients will answer a set of questions in a data collection sheet pertaining to

CONTACTS AND LOCATIONS:
Locations (1):
- American University of Beirut, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided